CLINICAL TRIAL: NCT06129539
Title: LIBELULA™: An Open-label, Single-arm, Multi-center, Phase 3 Study on the Efficacy, Safety, and Pharmacokinetics of Debio 4326, a Triptorelin 12-month Formulation, in Pediatric Participants With Central Precocious Puberty
Brief Title: A Study to Assess the Efficacy, Safety, and Pharmacokinetics of Debio 4326 in Pediatric Participants With Central Precocious Puberty (LIBELULA™ Clinical Trial)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Debiopharm International SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Debio 4326-301
Record Dates: First submitted 2023-11-08; First posted 2023-11-13 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Central Precocious Puberty
MeSH Terms: conditions — Puberty, Precocious

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Debio 4326 (Experimental): Participants will receive the first injection of Debio 4326, on Day 1 in Part A followed by a second injection 52 weeks later in Part B of the study.
  Interventions: Drug: Debio 4326

INTERVENTIONS:
Drug: Debio 4326 — Administered as an intramuscular (IM) injection

SUMMARY:
The primary objective of this study is to evaluate the efficacy of Debio 4326 in suppressing serum luteinizing hormone (LH) to prepubertal levels 52 weeks after the first Debio 4326 injection in pediatric participants with central precocious puberty (CPP).

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of central precocious puberty.
2. Onset of development of sex characteristics (i.e., breast development in girls or testicular enlargement in boys according to the Tanner method) before the age of 8 years in girls and 9 years in boys.
3. Initially, only participants aged (a) 5 to 8 years inclusive (i.e., <9 years) are eligible. The Sponsor will determine based on the recommendation of the DMC following the interim analysis whether participants aged (b) 2 to 4 years inclusive (i.e., <5 years) and/or (c) 9 to 10 years inclusive (i.e., <11 years) may be recruited.
4. Participant to receive at least 1 year of gonadotropin-releasing hormone agonist (GnRHa) therapy from study treatment start.
5. (a) Pre-treated participants: Start of initial GnRHa therapy no later than 18 months after onset of the first signs of CPP.

   (b) Treatment-naive participants: Start of Debio 4326 treatment no later than 18 months after onset of the first signs of CPP.
6. (a) Pre-treated participants: Difference between bone age (Greulich and Pyle method) and chronological age of ≥1 year based on historical values at the initiation of the GnRHa therapy.

   (b) Treatment-naive participants: Difference between bone age (Greulich and Pyle method) and chronological age of ≥1 year.
7. (a) Pre-treated participants: Pubertal-type LH response (LH ≥6 IU/L) following a GnRH/GnRHa stimulation test, or random non-stimulated serum LH >0.5 IU/L (if considered local standard of care), based on historical values prior to the initiation of GnRHa therapy.

   (b) Treatment-naive participants: Pubertal-type LH response (≥6 IU/L) 30 minutes following a GnRHa [leuprolide acetate 20 micrograms per kilogram (μg/kg) subcutaneous injection (SC)] stimulation test before treatment initiation.
8. (a) Pre-treated participants: Clinical evidence of puberty, defined as Tanner Staging ≥2 for breast development for girls and testicular volume ≥4 milliliter (mL) (cubic centimeter [cc]) for boys, prior to the initiation of GnRHa therapy.

   (b) Treatment-naive participants: Clinical evidence of puberty, defined as Tanner Staging ≥2 for breast development for girls and testicular volume ≥4 mL (cc) for boys.

Exclusion Criteria:

1. Gonadotropin-independent (peripheral) precocious puberty: gonadotropin-independent gonadal or adrenal sex steroid secretion.
2. (a) Pre-treated participants: Non-progressing, isolated premature thelarche prior to the initial GnRHa therapy.

   (b) Treatment-naive participants: Non-progressing, isolated premature thelarche.
3. Presence of an unstable intracranial tumor or an intracranial tumor potentially requiring neurosurgery or cerebral irradiation. Participants with hamartomas not requiring surgery are eligible.
4. Any other condition or chronic illness possibly interfering with growth (e.g., renal failure, diabetes, moderate to severe scoliosis, previously treated intracranial tumor).
5. Other than GnRHa therapy in pre-treated participants, any ongoing treatment with a potential effect on serum levels of gonadotropins or sex steroids, or possibly interfering with growth, opioids, central nervous system [CNS] stimulants).
6. Prior or current therapy with medroxyprogesterone acetate, growth hormone, or Insulin-like growth factor-1 (IGF-1).
7. Diagnosis of short stature, i.e., more than 2.25 standard deviations (SD) below the mean height-for-age.
8. Known history of seizures, epilepsy, and/or central nervous system disorders that may have been associated with seizures or convulsions.
9. Prior (within 2 months of study treatment start) or current use of medications that have been associated with seizures or convulsions.
10. Use of anticoagulants (heparin or coumarin derivatives).

Note: Other inclusion/exclusion criteria mentioned in the protocol may apply.

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Part A: Percentage of Participants With Suppression of Gonadotropin-Releasing Hormone Agonist Stimulated Serum Luteinizing Hormone (LH) to Less Than or Equal to (≤)5 International Units per Liter (IU/L) | Week 52 in Part A

SECONDARY OUTCOMES:
Parts A and B: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Adverse Events of Special Interest (AESIs) and Serious TEAEs | Up to 104 weeks
Parts A and B: Number of Participants with Clinically Significant Abnormalities in Vital Signs | Up to 104 weeks
Parts A and B: Change From Baseline in Body Weight | Up to 104 weeks
Parts A and B: Change From Baseline in Body Mass Index | Up to 104 weeks
Parts A and B: Number of Participants With Erythema, Swelling, and Induration at the Injection Site Immediately and 2 Hours After Each Debio 4326 Injection as per Investigator's Assessment | Up to 2 hours post-dose on Day 1 in both Parts A and B
Parts A and B: Number of Participants With Pain at the Injection Site Immediately and 2 Hours After Each Debio 4326 Injection as per Participant's Assessment Using the Wong-Baker FACES® Pain Rating Scale | Up to 2 hours post-dose on Day 1 in both Parts A and B
Parts A and B: Percentage of Participants Who do not Exhibit the Acute-on-Chronic (AOC) Phenomenon | Up to 48 hours post-dose on Day 3 in both Parts A and B
Parts A and B: Percentage of Participants With Stimulated Serum LH ≤5 IU/L | Up to Week 52 in both Parts A and B
Parts A and B: Percentage of Participants With Stimulated Serum LH ≤4 IU/L | Up to Week 52 in both Parts A and B
Parts A and B: Number of Participants With Change in Hormone Levels | Up to Week 52 in both Parts A and B
  The following hormones will be assessed: basal LH, follicle-stimulating hormone (FSH), estradiol, testosterone, GnRHa-stimulated LH, and GnRHa-stimulated FSH.
Parts A and B: Percentage of Girls With Prepubertal Serum Estradiol <20 pg/mL (<73 pmol/L) | Up to Week 52 in both Parts A and B
Parts A and B: Percentage of Boys With Testosterone <30 ng/dL (<1.0 nmol/L) | Up to Week 52 in both Parts A and B
Parts A and B: Change From Baseline in Height-for-Age Z Score | Baseline, up to Week 52 in both Parts A and B
Parts A and B: Number of Participants With Change From Baseline in Growth Velocity | Up to Week 52 in both Parts A and B
Percentage of Participants in Whom the Bone Age/Chronological Age Did Not Rise Relative to Baseline | Part A: Baseline, up to Week 52 in both Parts A and B
Parts A and B: Percentage of Participants Who Achieve Stabilization of Sexual Maturation (Regression or Stabilization Compared to Baseline by Tanner Staging) | Baseline, Weeks 26 and 52 in both Parts A and B
Parts A and B: Percentage of Girls With Regression of Uterine Length (Using Transabdominal Ultrasound) | Weeks 26 and 52 in both Parts A and B
Parts A and B: Percentage of Boys With Absence of Progression of Testis Volumes (Clinical Assessment With Orchidometer) | Weeks 26 and 52 in both Parts A and B
Parts A and B: Plasma Concentration of Triptorelin | Pre-dose and at multiple timepoints post-dose up to 52 weeks in Part A and 64 weeks in Part B
  The pharmacokinetics (PK) of triptorelin will be evaluated in plasma.
Percentage of Participants With Stimulated Serum LH Levels Greater Than (>)5 IU/L at Post Treatment Visit (PTV) | 64 weeks after the last Debio 4326 injection in Part A or B
  This outcome measure will be analyzed only in participants who stop all hormonal treatment with any GnRHa at end of treatment (EOT).
Part B: Accumulation Ratio on Maximum Serum Concentration (RacCmax) | At multiple timepoints post-dose up to 48 hours (Day 2) in Part B
Part B: Accumulation Ratio on Serum Concentration at the End of the Dosing Interval (RacCtrough) | At multiple timepoints post-dose up to 52 weeks in Part B

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Debiopharm International SA
Locations (31):
- United States (14):
  - TMC HealthCare, Tucson, Arizona
  - Rady Children's Hospital - San Diego, San Diego, California
  - University of California San Francisco-Benioff Children's Hospital, San Francisco, California
  - Wolfson's Children's Hospital, Jacksonville, Florida
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Indiana University/Riley Hospital for Children, Indianapolis, Indiana
  - University of Michigan, Ann Arbor, Michigan
  - Washington University, St Louis, Missouri
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Children's Hospital at Montefiore, New York, New York
  - Prisma Health Pediatric Endocrinology, Columbia, South Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas
  - Virginia Commonwealth University Health System, Richmond, Virginia
- Argentina (4):
  - Instituto de Investigaciones Metabolicas (IDIM), Buenos Aires
  - Centro Medico Dra Laura Maffei Investigacion Clinica Aplicada, Buenos Aires
  - Centro de Investigaciones Medicas Mar del Plata, Mar del Plata
  - Clinica Mayo de Urgencias Medicas Cruz Blanca S.R.L, San Miguel de Tucumán
- Brazil (10):
  - Hospital Da Criança de Brasília Jose Alencar, Brasília
  - CETI - Centro de Estudos em Terapias Inovadoras Ltda, Curitiba
  - Hospital Universitario Walter Cantidio, Fortaleza
  - Clínica de Endocrinologia e Metabologia Ltda, Lago Sul
  - Nucleo de Pesquisa Clínica do Rio Grande do Sul-NPCRS, Porto Alegre
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto, São José do Rio Preto
  - CPCLIN - Centro de Pesquisas Clínicas Ltda., São Paulo
  - CPQuali Pesquisa Clinica, São Paulo
  - Irmandade Santa Casa de São Paulo, São Paulo
  - Integral Pesquisa e Ensino, Votuporanga
- Chile (2):
  - ENDOMET, Antofagasta
  - Hospital Clinico San Borja Arriaran (HCSBA), Santiago
- Christus Latam Hub Center of Excellence and Innovation S C, Monterrey, Mexico

IPD SHARING:
Plan to Share IPD: No